CLINICAL TRIAL: NCT03636022
Title: Low-Cost, Virtual Reality System to Increase Access to Exposure Therapy for Anxiety and Obsessive Compulsive Disorders
Brief Title: Virtual Reality System for Anxiety and OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota HealthSolutions (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MinnesotaHealthSolutions; NCT03856567 (obsolete NCT alias)
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Obsessive-Compulsive Disorder
Keywords: Anxiety; OCD; Obsessive Compulsive Disorder; Generalized Anxiety Disorder; Social Phobia; Separation Anxiety; GAD; Youth; Teen; Therapy; Specific Phobia; Children
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder; Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation; Phobia, Specific

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to home exposure practice with or without the VR system, i.e., intervention or control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR System (Experimental): Participants will then be assigned one week of daily exposure homework. Patients randomized to the intervention condition will take home the VR system for homework.
  Interventions: Other: VR System
- Control Condition (Experimental): Participants will then be assigned one week of daily exposure homework. Participants assigned to control will be instructed to complete imaginal exposures.
  Interventions: Other: Control

INTERVENTIONS:
Other: VR System — Use of virtual reality to deliver exposure therapy
  Arms: VR System
Other: Control — Use of conventional delivery of exposure therapy
  Arms: Control Condition

SUMMARY:
Cognitive Behavioral Therapy with fear provoking exposures is the most effective therapy for anxiety disorders. The investigators aim to enhance this therapy with the use of virtual reality exposures. The human subjects study will test the effects of using VR for exposures compared to traditional imaginal exposures on anxiety symptom improvement, functioning, child engagement in an response to exposures, completion of exposure homework between treatment sessions, and length of treatment in weeks and length of treatment among children with anxiety disorders and/or obsessive compulsive disorder.

The funding award supports the development of the technology and the human subjects study. The subcontract to Mayo supports expert input to identify clinically relevant content for therapeutic videos on the VR system and the human subjects study to test the VR system.

DETAILED DESCRIPTION:
Seventy children with childhood anxiety disorders (CADs) or obsessive compulsive disorder (OCD) and a parent will be recruited to test the Phase II VR system with a randomized controlled mixed methods study. Participants will be identified through the Mayo Clinic Pediatric Anxiety Disorders Clinic (PADC). Participants will be randomly assigned to home exposure practice with or without the VR system, i.e., intervention or control, respectively. All participants in the study will participate in an introductory session in which participants complete two exposures related to content from their fear ladder, one with the VR system and analogous imaginal exposure. Each family will receive instructions for how to use the Mayo Clinic Anxiety Coach tablet app to record exposures during home practice. Participants will then be assigned one week of daily exposure homework for the intervention and control conditions. Participants randomized to the intervention condition will take home the VR system for homework completion and participants assigned to control will be instructed to complete imaginal exposures. One week after the introductory session, all participants will return for a session in which participants complete both types of exposure. Participants will also be assigned to a third generalization exposure, i.e., an exposure related to the baseline exposure that is higher on the fear ladder, to complete at their next anxiety clinic treatment sessions. SUDS ratings for each type of exposure will be recorded electronically via the Mayo Clinic Anxiety Coach. During the follow up session, an independent interviewer will observe participants' engagement during exposure and will interview participants and their parents about their experience with both types of exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7 to 17
2. Primary diagnosis of an anxiety disorder or obsessive compulsive disorder.

Exclusion Criteria:

1. History of and/or current diagnosis of: psychosis, autism, bipolar disorder, mental retardation, oppositional defiant disorder, PTSD, selective mutism or major depressive disorder.
2. Current sucidality or recent suicidal behavior.
3. Parent to be involved in study who is unable to adequately participate due to intellectual or psychiatric difficulties.
4. Starting or changing the dosage of psychiatric medications in the last 2 months.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Biggs, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available through the National Database for Clinical Trials Related to Mental Illness
Supporting Information: Study Protocol, ICF
Time Frame: 6 months following the study completion
Access Criteria: To be determined by the National Institute of Mental Health
URL: http://ndct.nimh.nih.gov

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VR System | Control Condition
Started | 25 | 20
Completed | 24 | 17
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VR System | Control Condition | Total
Number analyzed (Participants) | 25 | 20 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (2.6) | 13.1 (3.0) | 13.2 (2.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender at Birth: Female | 21 | 17 | 38
  Gender at Birth: Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Other | 1 | 0 | 1
  Race: Black | 1 | 1 | 2
  Race: Asian | 1 | 1 | 2
  Race: White | 22 | 18 | 40
Region of Enrollment [Number; unit: participants]
  United States | 25 | 20 | 45

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Subjective Units of Distress Scale (SUDS) at End of Session 1
Description: The SUDS - 0 to 10 ratings, where 0 indicates that participants feel no anxiety at all and 10 indicates that participants are experiencing maximum distress. The mean change in SUDS during the Session VR exposure versus mean change in SUDS during the conventional (control condition) verbal imaginal exposure.
Time Frame: Baseline and End of Session I, 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VR System | Control Condition
Number analyzed (Participants) | 24 | 17
units on a scale | -3.7 (2.0) | -3.6 (1.9)

2. Primary Outcome: Maximum SUDS Rating During Crossover Exposure
Description: Crossover exposure refers to the Session 2 virtual reality exposure for the control group and to the Session 2 imaginal exposure for the virtual reality group.
  The SUDs Rating Scale, or Subjective Units of Distress Scale (SUDs) is used to measure the intensity of distress or anxiety. The SUDs is a self-assessment tool rated on a scale from 0 to 10. Ten represents the highest level of distress and 0 represents no distress.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VR System | Control Condition
Number analyzed (Participants) | 24 | 17
units on a scale | 2.1 (2.3) | 2.5 (1.8)

3. Secondary Outcome: Homework Engagement
Description: Number of homework exposures completed.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: homework exposures completed
Arm/Group | VR System | Control Condition
Number analyzed (Participants) | 24 | 17
homework exposures completed | 5.4 (1.5) | 5.9 (1.3)

ADVERSE EVENTS:
Time Frame: Procedures for the present study occurred over two study sessions, each approximately 60-minutes and spaced a week apart. Data on adverse events were collected for each participant for their approximately one week of participation.
Arm/Group | VR System | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 0/25 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT03636022/Prot_SAP_000.pdf